CLINICAL TRIAL: NCT05035277
Title: AntiCoagulation Versus AcetylSalicylic Acid After Transcatheter Aortic Valve Implantation
Acronym: ACASA-TAVI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Øyvind Lie, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 247400; 2021-001554-61 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-09-05 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aortic Stenosis
Keywords: Transcatheter Aortic Valve Implantation; Transcatheter Aortic Valve Replacement; Antithrombotic therapy; Anticoagulation therapy; Antiplatelet therapy
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Aspirin; apixaban; Rivaroxaban; edoxaban

STUDY DESIGN:
Intervention Model Description: Parallel group prospective randomized open blinded endpoint (PROBE) trial
Who Masked: Outcomes Assessor
Masking Description: Separate endpoint adjudication committee blinded to randomized allocation of patients to treatment groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetylsalicylic acid (Active Comparator): Patients in the active control arm will receive 75 mg acetylsalicylic acid once daily indefinitely.
  Interventions: Drug: Acetylsalicylic acid
- Direct oral anticoagulation (DOAC) (Experimental): Patients in the experimental arm will receive an anti Xa-type DOAC (apixaban, rivaroxaban or edoxaban) in approved therapeutic dose for 12 months. The choice of DOAC agent will be made by the treating clinician after discussion with the patient. After 12 months, these patients will abort DOAC therapy. Acetylsalicylic acid, 75 mg once daily will be started after DOAC discontinuation and continued indefinitely.
  Interventions: Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban

INTERVENTIONS:
Drug: Acetylsalicylic acid — Acetylsalicylic acid 75 mg once daily is the current standard-of-care in TAVI patients without other indications for anticoagulation therapy.
  Other Names: B01A C06
  Arms: Acetylsalicylic acid
Drug: Apixaban — Standard dose apixaban will be one of the options for the patients in the experimental arm.
  Other Names: B01A F02
  Arms: Direct oral anticoagulation (DOAC)
Drug: Rivaroxaban — Standard dose rivaroxaban will be one of the options for the patients in the experimental arm.
  Other Names: B01A F01
  Arms: Direct oral anticoagulation (DOAC)
Drug: Edoxaban — Standard dose edoxaban will be one of the options for the patients in the experimental arm.
  Other Names: B01A F03
  Arms: Direct oral anticoagulation (DOAC)

SUMMARY:
ACASA-TAVI is a pragmatic randomized controlled trial assessing the value of anticoagulation therapy versus the standard antiplatelet therapy after transcatheter aortic valve implantation in patients with aortic stenosis. The trial will assess the efficacy of direct oral anticoagulation (DOAC) therapy compared to the standard single antiplatelet therapy to prevent degeneration of the valve and its safety in co-primary endpoints with blinded endpoint adjudication. The effect of DOAC therapy on hard clinical outcomes will be assessed during long-term follow-up.

DETAILED DESCRIPTION:
Aortic stenosis is a highly prevalent valvular disease and an important cause of morbidity and mortality in the elderly population. Transcatheter aortic valve implantation (TAVI) is an effective intervention in patients with severe aortic stenosis and low surgical risk. The procedure is highly effective, safe, and widely implemented. Current recommendations support transcatheter treatment of younger patients, including patients from 65 years of age with low surgical risk. This practice increases the importance of long-term valve maintenance.

Observational data have suggested that early signs of valve degeneration (i.e. hypo-attenuated leaflet thickening/thrombosis/reduced leaflet motion) are associated with an increased risk of embolic events. This is an increasing problem with emerging indications in younger populations. Because both ischemic and bleeding complications after TAVI can be life-threatening, it is important to establish the optimal anti-thrombotic treatment regime. Use of oral anticoagulation after implantation for bioprosthetic valves have been associated with resolved valve degeneration and possible favourable clinical effects.

The current practice guidelines recommend that oral anticoagulation may be considered for 3 months after open surgical bioprosthetic valve implantation. Patients with an independent indication for oral anticoagulation (i.e. atrial fibrillation or venous thromboembolism) are recommended to continue this treatment lifelong, but there is no recommendation for oral anticoagulation following TAVI in patients without other indications. In patients without indication for oral anticoagulation, the use of double anti-platelet therapy for 3-6 months following TAVI is recommended. However, single anti-platelet therapy with acetylsalicylic acid (ASA) without clopidogrel has been reported to improve bleeding outcomes and a composite of bleeding and ischemic outcomes. The effect of on oral anticoagulation-based treatment strategy compared to the standard single anti-platelet treatment strategy for valve maintenance after TAVI is unknown.

Increased anti-thrombotic treatment intensity may come at the cost of increased bleeding risk. Dual anti-platelet therapy and combination therapy with anticoagulation and anti-platelet therapy have both been associated with unfavourable outcomes. Combined anti-platelet and anti-coagulation treatment has been shown to reduce valve degeneration at the cost of increased bleeding. Conversely, single anti-platelet therapy and anti-coagulation with a direct oral anti-coagulant (DOAC) have been associated with similar bleeding risk. Bleeding rates in patients treated with anti-coagulation after TAVI have been reported to be slightly higher than in patients treated with ASA after TAVI, but patients with conventional indications for anti-coagulation have higher baseline bleeding risk than those without such indications. Therefore, the risk of bleeding in patients treated with DOAC or ASA following TAVI may be similar, but no randomized trials have been performed.

ACASA-TAVI will include 360 patients > 65 years and < 80 years of age who have undergone successful TAVI and have no conventional indication for DOAC in a prospective randomized open-label blinded-endpoint (PROBE) study. The intervention arm will be 12 month therapy with an anti-Xa type DOAC (without antiplatelet therapy) and the active control arm will be standard dose ASA. After 12 months, the intervention group will be switched to ASA maintenance. All patients will undergo clinical assessment, cardiac CT and echocardiography at 12 months with blinded endpoint adjudication by an independent committee.

Outcome measures will comply with the Valve Academic Research Consortium 3 (VARC-3) consensus, and are described in detail in the protocol. The co-primary endpoints at 12 months, hypo-attenuated leaflet thickening (HALT) and safety composite, must both be met for the trial to declare success.

The effect of the DOAC therapy on long-term major adverse cardiovascular events (MACE) will be assessed after 5 years and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Successful trans-catheter aortic valve implantation in patients aged >65 and <80 years old at the time of the procedure.

Exclusion Criteria:

* Strict indication for anticoagulation or anti-platelet drugs
* Strict contraindication for anticoagulation or anti-platelet drugs
* Overt cognitive failure
* Failure to obtain written informed consent
* Concomitant use of inducers or inhibitors of CYP3A4 or P-glycoprotein

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Hypo-attenuated leaflet thickening | 12 months
  First co-primary endpoint. The presence of hypo-attenuated leaflet thickening on dedicated cardiac CT after 12 months will be registered by a blinded expert reader. Intention-to-treat, superiority.
Safety composite - Incidence of Treatment Emergent Adverse Clinical Outcome | 12 months
  Second co-primary outcome. Composite of VARC-3 bleeding events, thromboembolic events (myocardial infarction or stroke) and all-cause mortality. Per-protocol, non-inferiority.
Major adverse cardiovascular events (MACE) | 5 years
  Primary outcome during long-term follow-up. The rate of the composite of Cardiac death, Aortic valve re-intervention, Stroke, Myocardial infarction, Heart failure hospitalization and Major, life-threatening, or disabling bleeding.
Major adverse cardiovascular events (MACE) | 10 years
  Primary outcome during long-term follow-up. The rate of the composite of Cardiac death, Aortic valve re-intervention, Stroke, Myocardial infarction, Heart failure hospitalization and Major, life-threatening, or disabling bleeding.

SECONDARY OUTCOMES:
Clinical efficacy | 12 months
  First hierarchical secondary outcome. Composite of of Freedom from all-cause mortality, Freedom from all stroke, Freedom from hospitalization for procedure- or valve-related causes, Freedom from KCCQ overall summary score <45 or decline from baseline of >10 points. Intention-to-treat, superiority.
Safety composite, superiority | 12 months
  Second hierarchical secondary outcome. Composite of VARC-3 bleeding events, thromboembolic events (myocardial infarction or stroke) and all-cause mortality. Same endpoint as second co-primary outcome, but intention-to-treat, superiority.
Thromboembolic events | 12 months
  Third hierarchical secondary outcome. Composite of myocardial infarction or stroke of any cause. Intention-to-treat population.
Bleeding events | 12 months
  Fourth hierarchical secondary outcome. Bleeding events according to VARC-3 definitions. Intention-to-treat population.
All-cause mortality | 12 months
  Fifth hierarchical secondary outcome. Intention-to-treat population.
The number of adverse events | 12 months
  First secondary safety endpoint. Safety population.
The number of serious adverse events | 12 months
  Second secondary safety endpoint. Safety population.
Life-threatening or disabling bleeding | 12 months
  Third secondary safety endpoint. Safety population. VARC-3 definition.
Major bleeding | 12 months
  Fourth secondary safety endpoint. Safety population. VARC-3 definition.
Minor bleeding | 12 months
  Fifth secondary safety endpoint. Safety population. VARC-3 definition.

OTHER OUTCOMES:
CT signs of valve degeneration | 12 months
  Exploratory outcome. Any evidence of reduced leaflet mobility, hypo-attenuated leaflet thickening or thrombus.
Echocardiographic signs of valve degeneration | 12 months
  Exploratory outcome. Change in transaortic pressure gradient assessed by echocardiography.
Cardiac function | 12 months
  Exploratory outcome. Change in left ventricular global longitudinal strain assessed by echocardiography.
Non-procedure-related life-threatening or disabling bleeding | 12 months
  Exploratory outcome. VARC-3 definition.
Number of major adverse clinical events | 12 months
  Exploratory outcome. Defined as stroke or transient ischemic attack of any cause, myocardial infarction, re-intervention on the aortic valve, death (cardiac, all-cause, non-cardiac) and heart failure hospitalization
Troponin T | 12 months
  Exploratory outcome. Assessment of blood samples.
N-terminal pro-B-type natriuretic peptide | 12 months
  Exploratory outcome. Assessment of blood samples.
Infective endocarditis | 12 months
  Exploratory outcome. Definition by Duke criteria.
Change in quality of life - Kansas City Cardiomyopathy Questionnaire | 12 months
  Exploratory outcome. Assessed by change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) score (score 0-100, Higher value indicates better quality of life).
Cognitive function | 12 months
  Exploratory outcome. Assessed by change in the Mini-cog score
Clinical efficacy | 5 years
  Composite of of Freedom from all-cause mortality, Freedom from all stroke, Freedom from hospitalization for procedure- or valve-related causes, Freedom from KCCQ overall summary score <45 or decline from baseline of >10 points. Intention-to-treat, superiority.
All-cause mortality | 5 years
  Fifth hierarchical secondary outcome. Intention-to-treat population.
Echocardiographic signs of valve degeneration | 5 years
  Exploratory outcome. Change in transaortic pressure gradient assessed by echocardiography.
Cardiac function | 5 years
  Exploratory outcome. Change in left ventricular global longitudinal strain assessed by echocardiography.
N-terminal pro-B-type natriuretic peptide | 5 years
  Exploratory outcome. Assessment of blood samples.
Troponin T | 5 years
  Exploratory outcome. Assessment of blood samples.
Individual components of MACE | 5 years
  Exploratory outcome. Assessment of the individual components of MACE (the primary outcome at long-term follow-up).
Change in quality of life - Kansas City Cardiomyopathy Questionnaire | 5 years
  Exploratory outcome. Assessed by change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) score (score 0-100, Higher value indicates better quality of life).
Cognitive function | 5 years
  Exploratory outcome. Assessed by change in the Mini-cog score
Infective endocarditis | 5 years
  Exploratory outcome. Definition by Duke criteria.
Clinical efficacy | 10 years
  Composite of of Freedom from all-cause mortality, Freedom from all stroke, Freedom from hospitalization for procedure- or valve-related causes, Freedom from KCCQ overall summary score <45 or decline from baseline of >10 points. Intention-to-treat, superiority.
All-cause mortality | 10 years
  Fifth hierarchical secondary outcome. Intention-to-treat population.
Echocardiographic signs of valve degeneration | 10 years
  Exploratory outcome. Change in transaortic pressure gradient assessed by echocardiography.
Cardiac function | 10 years
  Exploratory outcome. Change in left ventricular global longitudinal strain assessed by echocardiography.
N-terminal pro-B-type natriuretic peptide | 10 years
  Exploratory outcome. Assessment of blood samples.
Troponin T | 10 years
  Exploratory outcome. Assessment of blood samples.
Individual components of MACE | 10 years
  Exploratory outcome. Assessment of the individual components of MACE (the primary outcome at long-term follow-up).
Change in quality of life - Kansas City Cardiomyopathy Questionnaire | 10 years
  Exploratory outcome. Assessed by change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) score (score 0-100, Higher value indicates better quality of life).
Cognitive function | 10 years
  Exploratory outcome. Assessed by change in the Mini-cog score
Infective endocarditis | 10 years
  Exploratory outcome. Definition by Duke criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind H Lie, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo Univesity Hospital - Ullevål, Oslo
  - Oslo University Hospital - Rikshospitalet, Oslo

IPD SHARING:
Plan to Share IPD: Yes
The application to share IPD is pending with the ethical committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be made available with the publication of the primary analysis and remain available for 1 year. Thereafter, it can be made available upon request.
Access Criteria: Researchers and clinicians with valid medical questions to be addressed. The data will not be available for commercial use.

REFERENCES:
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579
- [Derived] Dodgson CS, Beitnes JO, Klove SF, Herstad J, Opdahl A, Undseth R, Eek CH, Broch K, Gullestad L, Aaberge L, Lunde K, Bendz B, Lie OH. An investigator-sponsored pragmatic randomized controlled trial of AntiCoagulation vs AcetylSalicylic Acid after Transcatheter Aortic Valve Implantation: Rationale and design of ACASA-TAVI. Am Heart J. 2023 Nov;265:225-232. doi: 10.1016/j.ahj.2023.08.010. Epub 2023 Aug 25. PMID 37634655

DOCUMENTS (1):
  • Study Protocol (2022-02-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT05035277/Prot_002.pdf